CLINICAL TRIAL: NCT00501228
Title: RhG-CSF (Filgrastim) Treatment of Severe Epithelial/Endothelial or Solid Organ-Specific Tissue Damage In Stem Cell Transplant Recipients
Brief Title: Tissue Repair in Stem Cell Transplant Recipients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID02-300
Record Dates: First submitted 2007-07-12; First posted 2007-07-16 (Estimated); Results first posted 2009-11-20 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-07

CONDITIONS: Graft-Versus-Host Disease
Keywords: Graft-Versus-Host Disease; Stem Cell Transplantation; Tissue Repair; Organ-Specific Tissue Damage; Filgrastim; RhG-CSF
MeSH Terms: conditions — Graft vs Host Disease | interventions — Filgrastim; pegylated granulocyte colony-stimulating factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Filgrastim Injections (Experimental)
  Interventions: Drug: Filgrastim

INTERVENTIONS:
Drug: Filgrastim — 5 mg/kg ID Once Daily x 1 Week
  Other Names: RhG-CSF

SUMMARY:
Primary Objective:

1. To determine whether rhG-CSF treatment will increase the frequency of donor-derived cells contributing to repair of damaged epithelial/endothelial or solid organ-specific tissue caused by graft-versus-host disease (GVHD) in patients who underwent sex-mismatched stem cell transplantation.

Secondary Objective:

1. To determine whether rhG-CSF treatment can alleviate GVHD-induced damage to epithelial/endothelial or solid organ-specific tissue.

DETAILED DESCRIPTION:
It has been found that cells circulating in the blood are capable of forming cells lining the oral cavity, skin cells, and/or cells of various organs. RhG-CSF is used to support cell recovery after stem cell transplantation and is commercially available.

Before treatment starts, participants will have at least one (and up to three) biopsy(ies) of damaged tissue performed to find out about the severity of tissue damage. A biopsy is taken with a large needle. Women able to have children must have a negative blood pregnancy test.

Participants in this study will receive rhG-CSF as an injection under the skin once a day over one week. This will be repeated every other week for a total of 4 weeks. Blood tests (about 2 teaspoons each) will be performed 3 times while at M. D. Anderson or once a week while outpatient to make sure that the white blood count stays in a safe range. Participants will have at least one (and up to three) biopsy(ies) again performed about 8 weeks after the start of rhG-CSF treatment. An additional biopsy at 3 months after the start rhG-CSF treatment will only be performed in case your regular treatment follow up requires it, and not for research purposes only.

Participants will be taken off study if severe side effects occur. The study will end after the last biopsy or biopsies are taken, about 3 months after the start of rhG-CSF treatment.

This is an investigational study. RhG-CSF is FDA approved and commercially available, though its use in this study is investigational. A maximum of 5 patients will be treated on this protocol. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who underwent allogeneic bone marrow or peripheral blood stem cell transplantation.
2. Patients should have engrafted with WBC concentration >3000/ul. Patients should have acute GVHD overall > grade 2 or chronic GVHD.
3. Patients with acute GVHD or chronic GVHD including patients refractory to steroid treatment.
4. Donors and patients must be of different gender.
5. Patients must sign an informed consent indicating that they are aware of the investigational nature of this study in keeping with the policies of the hospital.
6. The only acceptable consent form is the one attached at the end of this protocol.
7. Patients agree to biopsy tissue areas unaffected by GVHD for only research purposes.

Exclusion Criteria:

1. Patients who are allergic to rhG-CSF.
2. Patients who had any prior allogeneic stem cell transplantation using a sex mismatched donor other than the donor used for the previous stem cell allotransplantation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2003-02; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin J. Korbling, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 06/15/2005 through 05/03/2006. All participants enrolled at U.T. M.D. Anderson Cancer Center.
Pre-assignment Details: Study terminated early due to lack of accrual.
Period: Overall Study
Arm/Group | Filgrastim Injections
Started | 2
Completed | 1
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Filgrastim Injections
Number analyzed (Participants) | 2
Age Continuous [Median (Full Range); unit: years] | 48 [40 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Donor Derived Cells After G-CSF Therapy
Description: In each patient, the number of donor derived (dd) cells in solid organ tissue specimens measured by biopsy of relevant tissue at initiation of rhG-CSF treatment (baseline) and at eight weeks post allogeneic transplant.
Time Frame: Baseline + 8 Weeks post transplant
Population: No analysis was done. Only one eligible patient was able to complete treatment.
Arm/Group | Filgrastim Injections
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Filgrastim Injections
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

LIMITATIONS AND CAVEATS:
Study was closed because of the very limited number of patients enrolled. Patients eligible for enrollment were not willing to undergo 4 weekly cycles of G-CSF treatment because of the well known side effect of bone pain.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No